CLINICAL TRIAL: NCT05013671
Title: Benign Paroxysmal Positional Vertigo (BPPV) in Nursing Homes: Treatment Efficacy and Impact on Balance, Gait and Falls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, JSpildooren, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BPPV in WCZ - 001
Record Dates: First submitted 2020-09-17; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: BPPV
Keywords: Benign Paroxysmal Positional Vertigo; vertigo; older adults; frailty; nursing home
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Frailty

STUDY DESIGN:
Intervention Model Description: First, the nursing home resident will be assessed for the presence of BPPV. Based on the presence of BPPV, two groups will be formed: BPPV-group and control group. The residents suffering from BPPV will undergo balance tests and will be treated for their BPPV (BPPV-group). The nursing home residents with BPPV will be matched to residents without the disease (case control design) and will also undergo balance tests. At 1,3,6 and 12 months the presence of balance problems will be followed up in both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- residents with BPPV (Active Comparator)
  Interventions: Other: repositioning maneuvers; Other: balance
- residents without BPPV (Other)
  Interventions: Other: balance

INTERVENTIONS:
Other: repositioning maneuvers — The calcium crystals floating in the endolymphatic fluid will put back in place by putting the patient in several sitting and lying positions during specific repositioning maneuvers. During these maneuvers the calcium crystals will float from the semicircular canals back into the utriculus, after which the dizziness symptoms should disappear
  Arms: residents with BPPV
Other: balance — compare the balance of residents with BPPV with residents without BPPV

SUMMARY:
BPPV is a benign condition of the balance organ, localized in the inner ear, in which calcium crystals loosen up and move freely in the endolymphatic fluid of the inner ear (more specifically in the semi-circular canals). During certain posture changes or head movements, these moving calcium crystals cause dizziness and balance problems. The general objective of the study is to evaluate the impact of BPPV on the balance of older adults in nursing homes. For this purpose, we will compare the balance of residents with BPPV with residents without BPPV. Furthermore, we will identify the impact of treatment on balance problems and fall risk in older adults in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized for at least 3 months
* Willing to participate
* Able to understand simple instructions
* Able to stand independently for 10 seconds (with the use of a walking aid)

Exclusion Criteria:

* Diagnosis of progressive neurological conditions resulting in a fast deterioration (i.e. amyotrophic lateral sclerosis or residents with palliative care)
* Participation in a rehabilitation program at the current time for a pathology of less than 6 months
* Contra-indication for vestibular testing such as heart failure or fear

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The presence of BPPV | Baseline
  This will be measured using the side lying test (posterior and anterior canal BPPV) and the side lying test for horizontal canal BPPV.
The presence of BPPV | Month 1
  This will be measured using the side lying test (posterior and anterior canal BPPV) and the side lying test for horizontal canal BPPV.
The presence of BPPV | Month 3
  This will be measured using the side lying test (posterior and anterior canal BPPV) and the side lying test for horizontal canal BPPV.
The presence of BPPV | Month 6
  This will be measured using the side lying test (posterior and anterior canal BPPV) and the side lying test for horizontal canal BPPV.
The presence of BPPV | Month 12
  This will be measured using the side lying test (posterior and anterior canal BPPV) and the side lying test for horizontal canal BPPV.
Dizziness Handicap Inventory | Baseline
  Self-reported impact of dizziness on daily life. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0. The higher score, the greater the perceived handicap due to dizziness.
Dizziness Handicap Inventory | Month 1
  Self-reported impact of dizziness on daily life. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0. The higher score, the greater the perceived handicap due to dizziness.
Dizziness Handicap Inventory | Month 3
  Self-reported impact of dizziness on daily life. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0. The higher score, the greater the perceived handicap due to dizziness.
Dizziness Handicap Inventory | Month 6
  Self-reported impact of dizziness on daily life. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0. The higher score, the greater the perceived handicap due to dizziness.
Dizziness Handicap Inventory | Month 12
  Self-reported impact of dizziness on daily life. There is a maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) and a minimum score of 0. The higher score, the greater the perceived handicap due to dizziness.
Falls Efficacy Scale International | Baseline
  Measuring fear of falling during daily and social activities. There is a minimum score of 16 (no concern about falling) to maximum 64 (severe concern about falling).
Falls Efficacy Scale International | Month 1
  Measuring fear of falling during daily and social activities. There is a minimum score of 16 (no concern about falling) to maximum 64 (severe concern about falling).
Falls Efficacy Scale International | Month 3
  Measuring fear of falling during daily and social activities. There is a minimum score of 16 (no concern about falling) to maximum 64 (severe concern about falling).
Falls Efficacy Scale International | Month 6
  Measuring fear of falling during daily and social activities. There is a minimum score of 16 (no concern about falling) to maximum 64 (severe concern about falling).
Falls Efficacy Scale International | Month 12
  Measuring fear of falling during daily and social activities. There is a minimum score of 16 (no concern about falling) to maximum 64 (severe concern about falling).
Static balance | Baseline
  Measuring balance in four positions: stand straight with eyes open (firm surface), standing straight with eyes closed (firm surface), standing straight on a foam with eyes open and standing straight on a foam with eyes closed.
Static balance | Month 1
  Measuring balance in four positions: stand straight with eyes open (firm surface), standing straight with eyes closed (firm surface), standing straight on a foam with eyes open and standing straight on a foam with eyes closed.
Static balance | Month 3
  Measuring balance in four positions: stand straight with eyes open (firm surface), standing straight with eyes closed (firm surface), standing straight on a foam with eyes open and standing straight on a foam with eyes closed.
Static balance | Month 6
  Measuring balance in four positions: stand straight with eyes open (firm surface), standing straight with eyes closed (firm surface), standing straight on a foam with eyes open and standing straight on a foam with eyes closed.
Static balance | Month 12
  Measuring balance in four positions: stand straight with eyes open (firm surface), standing straight with eyes closed (firm surface), standing straight on a foam with eyes open and standing straight on a foam with eyes closed.
Timed up and Go (TUG) | Baseline
  Measuring dynamic balance and gait during TUG over a 3 meter distance
Timed up and Go (TUG) | Month 1
  Measuring dynamic balance and gait during TUG over a 3 meter distance
Timed up and Go (TUG) | Month 3
  Measuring dynamic balance and gait during TUG over a 3 meter distance
Timed up and Go (TUG) | Month 6
  Measuring dynamic balance and gait during TUG over a 3 meter distance
Timed up and Go (TUG) | Month 12
  Measuring dynamic balance and gait during TUG over a 3 meter distance
360° turn | Baseline
  Measuring dynamic balance during a 360° turn
360° turn | month 1
  Measuring dynamic balance during a 360° turn
360° turn | month 3
  Measuring dynamic balance during a 360° turn
360° turn | month 6
  Measuring dynamic balance during a 360° turn
360° turn | month 12
  Measuring dynamic balance during a 360° turn
10 meter walk test | Baseline
  The participant walks 10 meters at a comfortable pace. A walking aid/orthosis can be used during the test, but the help from a third party during is prohibited. Body movements will be registered wuth the use of ADPM sensors.
10 meter walk test | Month 1
  The participant walks 10 meters at a comfortable pace. A walking aid/orthosis can be used during the test, but the help from a third party during is prohibited. Body movements will be registered wuth the use of ADPM sensors.
10 meter walk test | Month 3
  The participant walks 10 meters at a comfortable pace. A walking aid/orthosis can be used during the test, but the help from a third party during is prohibited. Body movements will be registered wuth the use of ADPM sensors.
10 meter walk test | Month 6
  The participant walks 10 meters at a comfortable pace. A walking aid/orthosis can be used during the test, but the help from a third party during is prohibited. Body movements will be registered wuth the use of ADPM sensors.
10 meter walk test | Month 12
  The participant walks 10 meters at a comfortable pace. A walking aid/orthosis can be used during the test, but the help from a third party during is prohibited. Body movements will be registered wuth the use of ADPM sensors.
Knee extensor strength | Baseline
  The strength of the knee extensor muscles of the right leg will be assessed with hand-held dynamometry (MicroFET). This dynamometer is placed between the leg segment to be evaluated and the examiner's hand. Participants were asked to sit with their legs over the end of a standard, examination table, with hips and knees flexed to 90. Participants have to hold the side-edges of the table with their hands and carry out a maximal isometric voluntary contraction for 3-5 s. The break method will be used to asses the knee extensor strength. This test will be performed 3 times.
Knee extensor strength | Month 1
  The strength of the knee extensor muscles of the right leg will be assessed with hand-held dynamometry (MicroFET). This dynamometer is placed between the leg segment to be evaluated and the examiner's hand. Participants were asked to sit with their legs over the end of a standard, examination table, with hips and knees flexed to 90. Participants have to hold the side-edges of the table with their hands and carry out a maximal isometric voluntary contraction for 3-5 s. The break method will be used to asses the knee extensor strength. This test will be performed 3 times.
Knee extensor strength | Month 3
  The strength of the knee extensor muscles of the right leg will be assessed with hand-held dynamometry (MicroFET). This dynamometer is placed between the leg segment to be evaluated and the examiner's hand. Participants were asked to sit with their legs over the end of a standard, examination table, with hips and knees flexed to 90. Participants have to hold the side-edges of the table with their hands and carry out a maximal isometric voluntary contraction for 3-5 s. The break method will be used to asses the knee extensor strength. This test will be performed 3 times.
Knee extensor strength | Month 6
  The strength of the knee extensor muscles of the right leg will be assessed with hand-held dynamometry (MicroFET). This dynamometer is placed between the leg segment to be evaluated and the examiner's hand. Participants were asked to sit with their legs over the end of a standard, examination table, with hips and knees flexed to 90. Participants have to hold the side-edges of the table with their hands and carry out a maximal isometric voluntary contraction for 3-5 s. The break method will be used to asses the knee extensor strength. This test will be performed 3 times.
Knee extensor strength | Month 12
  The strength of the knee extensor muscles of the right leg will be assessed with hand-held dynamometry (MicroFET). This dynamometer is placed between the leg segment to be evaluated and the examiner's hand. Participants were asked to sit with their legs over the end of a standard, examination table, with hips and knees flexed to 90. Participants have to hold the side-edges of the table with their hands and carry out a maximal isometric voluntary contraction for 3-5 s. The break method will be used to asses the knee extensor strength. This test will be performed 3 times.

SECONDARY OUTCOMES:
Fall incidents | Baseline
  Falls incidents retrieved from nursing home staff
Fall incidents | month 1
  Falls incidents retrieved from nursing home staff
Fall incidents | month 3
  Falls incidents retrieved from nursing home staff
Fall incidents | month 6
  Falls incidents retrieved from nursing home staff
Fall incidents | month 12
  Falls incidents retrieved from nursing home staff
Katz-ADL (retrospective data retrieved from patient files) | Baseline
  The Katz-scale assesses functional status as a measurement of the client's ability to perform activities of daily living independently. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Katz-ADL (retrospective data retrieved from patient files) | Month 1
  The Katz-scale assesses functional status as a measurement of the client's ability to perform activities of daily living independently. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Katz-ADL (retrospective data retrieved from patient files) | Month 3
  The Katz-scale assesses functional status as a measurement of the client's ability to perform activities of daily living independently. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Katz-ADL (retrospective data retrieved from patient files) | Month 6
  The Katz-scale assesses functional status as a measurement of the client's ability to perform activities of daily living independently. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Katz-ADL (retrospective data retrieved from patient files) | Month 12
  The Katz-scale assesses functional status as a measurement of the client's ability to perform activities of daily living independently. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Medication (retrospective data retrieved from patient files) | Baseline
  Medication that may affect the vestibular system will be retrieved from patient files.
Medication (retrospective data retrieved from patient files) | Month 1
  Medication that may affect the vestibular system will be retrieved from patient files.
Medication (retrospective data retrieved from patient files) | Month 3
  Medication that may affect the vestibular system will be retrieved from patient files.
Medication (retrospective data retrieved from patient files) | Month 6
  Medication that may affect the vestibular system will be retrieved from patient files.
Medication (retrospective data retrieved from patient files) | Month 12
  Medication that may affect the vestibular system will be retrieved from patient files.
Sleep pattern (retrospective data retrieved from patient files) | Baseline
  If the participant has a normal/disturbed sleep pattern.
Sleep pattern (retrospective data retrieved from patient files) | Month 1
  If the participant has a normal/disturbed sleep pattern.
Sleep pattern (retrospective data retrieved from patient files) | Month 3
  If the participant has a normal/disturbed sleep pattern.
Sleep pattern (retrospective data retrieved from patient files) | Month 6
  If the participant has a normal/disturbed sleep pattern.
Sleep pattern (retrospective data retrieved from patient files) | Month 12
  If the participant has a normal/disturbed sleep pattern.
Comorbidities (retrospective data retrieved from patient files) | Baseline
  The number and kind of comorbidities including COVID-19 infection in the participants history.
Comorbidities (retrospective data retrieved from patient files) | Month 1
  The number and kind of comorbidities including COVID-19 infection in the participants history.
Comorbidities (retrospective data retrieved from patient files) | Month 3
  The number and kind of comorbidities including COVID-19 infection in the participants history.
Comorbidities (retrospective data retrieved from patient files) | Month 6
  The number and kind of comorbidities including COVID-19 infection in the participants history.
Comorbidities (retrospective data retrieved from patient files) | Month 12
  The number and kind of comorbidities including COVID-19 infection in the participants history.
Nutrition (retrospective data retrieved from patient files) | Baseline
  If the participant is on a specific diet (i.e.salt-free diet, low fat diet, calcium-rich diet etc.) and if there is a loss of apetite.
Nutrition (retrospective data retrieved from patient files) | Month 1
  If the participant is on a specific diet (i.e.salt-free diet, low fat diet, calcium-rich diet etc.) and if there is a loss of apetite.
Nutrition (retrospective data retrieved from patient files) | Month 3
  If the participant is on a specific diet (i.e.salt-free diet, low fat diet, calcium-rich diet etc.) and if there is a loss of apetite.
Nutrition (retrospective data retrieved from patient files) | Month 6
  If the participant is on a specific diet (i.e.salt-free diet, low fat diet, calcium-rich diet etc.) and if there is a loss of apetite
Nutrition (retrospective data retrieved from patient files) | Month 12
  If the participant is on a specific diet (i.e.salt-free diet, low fat diet, calcium-rich diet etc.) and if there is a loss of apetite.
Geriatric Depression Scale (GDS) | Baseline
  The GDS is commonly used as a routine part of a Comprehensive Geriatric Assessment. One point is assigned to each answer and the cumulative score is rated on a scoring grid.[2] The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".
Geriatric Depression Scale (GDS) | Month 1
  The GDS is commonly used as a routine part of a Comprehensive Geriatric Assessment. One point is assigned to each answer and the cumulative score is rated on a scoring grid.[2] The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".
Geriatric Depression Scale (GDS) | Month 3
  The GDS is commonly used as a routine part of a Comprehensive Geriatric Assessment. One point is assigned to each answer and the cumulative score is rated on a scoring grid.[2] The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".
Geriatric Depression Scale (GDS) | Month 6
  The GDS is commonly used as a routine part of a Comprehensive Geriatric Assessment. One point is assigned to each answer and the cumulative score is rated on a scoring grid.[2] The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".
Geriatric Depression Scale (GDS) | Month 12
  The GDS is commonly used as a routine part of a Comprehensive Geriatric Assessment. One point is assigned to each answer and the cumulative score is rated on a scoring grid.[2] The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".
Montreal Cognitive Assessment (MOCA) | Baseline
  The Montreal Cognitive Assessment (MoCA) is a brief 30-question test that takes around 10 to 12 minutes to complete and helps assess people for dementia.
Montreal Cognitive Assessment (MOCA) | Month 1
  The Montreal Cognitive Assessment (MoCA) is a brief 30-question test that takes around 10 to 12 minutes to complete and helps assess people for dementia.
Montreal Cognitive Assessment (MOCA) | Month 3
  The Montreal Cognitive Assessment (MoCA) is a brief 30-question test that takes around 10 to 12 minutes to complete and helps assess people for dementia.
Montreal Cognitive Assessment (MOCA) | Month 6
  The Montreal Cognitive Assessment (MoCA) is a brief 30-question test that takes around 10 to 12 minutes to complete and helps assess people for dementia.
Montreal Cognitive Assessment (MOCA) | Month 12
  The Montreal Cognitive Assessment (MoCA) is a brief 30-question test that takes around 10 to 12 minutes to complete and helps assess people for dementia.
Hospital anxiety and depression scale (HADS) | Baseline
  The Hospital Anxiety and Depression Scale (HADS) is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients. Only the questions related to the anxiety subscale will be used. The total score ranges from 0 to 21, a score >8 denotes anxiety.
Hospital anxiety and depression scale (HADS) | Month 1
  The Hospital Anxiety and Depression Scale (HADS) is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients. Only the questions related to the anxiety subscale will be used. The total score ranges from 0 to 21, a score >8 denotes anxiety.
Hospital anxiety and depression scale (HADS) | Month 3
  The Hospital Anxiety and Depression Scale (HADS) is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients. Only the questions related to the anxiety subscale will be used. The total score ranges from 0 to 21, a score >8 denotes anxiety.
Hospital anxiety and depression scale (HADS) | Month 6
  The Hospital Anxiety and Depression Scale (HADS) is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients. Only the questions related to the anxiety subscale will be used. The total score ranges from 0 to 21, a score >8 denotes anxiety.
Hospital anxiety and depression scale (HADS) | Month 12
  The Hospital Anxiety and Depression Scale (HADS) is a frequently used self-rating scale developed to assess psychological distress in non-psychiatric patients. Only the questions related to the anxiety subscale will be used. The total score ranges from 0 to 21, a score >8 denotes anxiety.
Frailty status | Baseline
  Frailty status using Fried Criteria
Frailty status | month 1
  Frailty status using Fried Criteria
Frailty status | month 3
  Frailty status using Fried Criteria
Frailty status | month 6
  Frailty status using Fried Criteria
Frailty status | month 12
  Frailty status using Fried Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Joke Spildooren, prof. dr., Principal Investigator — Hasselt University; Laura Casters, drs., Study Chair — Hasselt University
Locations (1):
- WZC Leopoldspark, Leopoldsburg, Belgium